CLINICAL TRIAL: NCT03237988
Title: A Phase 1, Open-label, Randomized, Single-dose, Three-way Crossover Study to Evaluate the Pharmacokinetics of a New Tablet Formulation of CPI-444 in Fed and Fasted Healthy Male and Female Subjects
Brief Title: Study to Evaluate the Pharmacokinetics of a New Tablet Formulation of CPI-444 in Fed and Fasted Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CPI-444-002
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ciforadenant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence ABC (Active Comparator): 100 mg CPI-444, given orally as a 1 × 100-mg capsule, after an overnight fast of at least 10 hours (fasted); 100 mg CPI-444, given orally as a 1 × 100-mg tablet, after an overnight fast of at least 10 hours (fasted); 100 mg CPI-444, given orally as a 1 × 100-mg tablet, 30 minutes after the start of a high-fat breakfast (fed).
  Interventions: Drug: CPI-444 Capsules; Drug: CPI-444 Tablets
- Sequence BCA (Active Comparator): 100 mg CPI-444, given orally as a 1 × 100-mg tablet, after an overnight fast of at least 10 hours (fasted); 100 mg CPI-444, given orally as a 1 × 100-mg tablet, 30 minutes after the start of a high-fat breakfast (fed); 100 mg CPI-444, given orally as a 1 × 100-mg capsule, after an overnight fast of at least 10 hours (fasted).
  Interventions: Drug: CPI-444 Capsules; Drug: CPI-444 Tablets
- Sequence CAB (Active Comparator): 100 mg CPI-444, given orally as a 1 × 100-mg tablet, 30 minutes after the start of a high-fat breakfast (fed); 100 mg CPI-444, given orally as a 1 × 100-mg capsule, after an overnight fast of at least 10 hours (fasted); 100 mg CPI-444, given orally as a 1 × 100-mg tablet, after an overnight fast of at least 10 hours (fasted).
  Interventions: Drug: CPI-444 Capsules; Drug: CPI-444 Tablets

INTERVENTIONS:
Drug: CPI-444 Capsules — 100mg Capsule
Drug: CPI-444 Tablets — 100mg Tablets

SUMMARY:
This will be a Phase 1, open-label, randomized, 3-way crossover study to evaluate PK, safety, and tolerability of a new tablet formulation of CPI-444 and to evaluate the effect of food on single oral doses of CPI-444 tablets in healthy male and female subjects. Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the first dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, 18 to 65 years of age, inclusive, at Screening.
2. Body mass index between 18.5 and 32.0 kg/m2, inclusive, at Screening.
3. In good health.
4. Females will be nonpregnant and nonlactating, and females of childbearing potential and males will agree to use contraception.
5. Able to comprehend and willing to sign an Informed Consent Form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder.
2. Subjects who have received any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose.
3. Females of childbearing potential who are pregnant or lactating. Females of non-childbearing potential are defined as permanently sterile or postmenopausal. Postmenopausal status will be confirmed with a screening serum follicle-stimulating hormone (FSH) level greater than 40 mIU/mL.
4. A history or evidence of clinically significant gastrointestinal disease, including ulcers, gastro-esophageal reflux disease, or gastritis.
5. A history of alcoholism or drug/chemical abuse within 2 years prior to Period 1 Check-in.
6. Regular alcohol consumption of >21 units per week for males and >14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
7. Positive urine drug screen (confirmed by repeat) at Screening (does not include alcohol) or Check-in (does include alcohol).
8. Use of prescription or nonprescription drugs, including vitamins, herbal, and dietary supplements (ie, St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of IMP.
9. Use of tobacco, smoking cessation products, or products containing nicotine (including, but not limited to, cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine lozenges, or nicotine gum) within 6 months prior to Period 1 Check-in until Discharge from the CRU following the final dose.
10. Consumption of foods and beverages containing poppy seeds, grapefruit, or Seville oranges will not be allowed from 7 days prior to Period 1 Check-in until Discharge from the CRU following the final dose.
11. Consumption of caffeine-containing foods and beverages will not be allowed from 72 hours prior to Check-in until Discharge on Day 4 of each treatment period.
12. Poor peripheral venous access.
13. Evidence of renal impairment at Screening, as indicated by an estimated creatinine clearance of less than 80 mL/min using the Cockcroft-Gault equation.
14. Screening chemistry laboratory values as follows: gamma-glutamyltransferase, aspartate aminotransferase, and ALT >1.5 × institutional upper limit of normal (ULN), total bilirubin >1.5 × institutional ULN.
15. A history of seizures (not including simple febrile seizures in childhood);
16. Multiple drug allergies or allergies to any of the components of CPI-444 tablets or CPI 444 resinate capsules.
17. Known history of human immunodeficiency virus or active infection requiring therapy, or positive tests for hepatitis B surface antigen or hepatitis C antibody.
18. Any vaccination against infectious diseases (ie, influenza, varicella) within 28 days of first dose.
19. Donation or loss of greater than 400 mL of blood from 2 months prior to Screening, donation of platelets from 6 weeks prior to Screening, or plasma from 2 weeks prior to Screening through the Follow-up phone call.
20. Receipt of blood products within 2 months prior to Period 1 Check-in.
21. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
AUC0-∞: AUC from time zero to infinity | Predose through 72 hours postdose
  Area under the plasma concentration-time curve (AUC) from time zero to infinity
AUC0-tz: AUC from time zero to last quantifiable concentration | Predose through 72 hours postdose
  AUC from time zero to the last quantifiable concentration
%AUCex: Percentage of AUC0-∞ that was due to extrapolation from the last quantifiable concentration to infinity | Predose through 72 hours postdose
  Percentage of AUC0-∞ that was due to extrapolation from the last quantifiable concentration to infinity

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No